CLINICAL TRIAL: NCT04808492
Title: The Effects of CureWave Laser on Paraspinal Muscle Oxygenation, Pressure Pain Thresholds, Muscle Edema, Muscle Quality, and Perceived Outcomes in Patients With Chronic Low Back Pain.
Brief Title: The Effect of High Intensity Laser on Muscle Quality and Pain in Those With Low Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: University of Central Florida (Other)
Collaborators: Curewave Laser, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001355
Record Dates: First submitted 2021-03-04; First posted 2021-03-22 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Low Back Pain
Keywords: low back pain; Laser; Perceived Pain; Perceived Disability
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participating subjects will be blinded to group assignment. Also, the outcomes assessor analyzing the data will be blinded to group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CureWave High Intensity Laser (Experimental): The participant will lie prone and the HILT will be administered in two preliminary test locations. In order to evaluate any possible adverse reactions, the initial treatment location will be delivered at a decreased intensity at two separate locations above the target treatment areas. The Power for these two locations will be at a half dose (22 W) for one minute each. The initial, half dose treatment area is indicated by the Blue circles in the image below. Upon conclusion of the initial test treatments (at half dose), the skin with be evaluated for excessive redness or any other changes in skin appearance. Also, the participant will be asked about any discomfort. Should no unanticipated changes in skin appearance occur and the participant reports no discomfort, the treatment will be administered. The process of applying the laser at half dosage will occur prior to each treatment.
  Interventions: Device: CureWave High Intensity Laser
- Control (Placebo Comparator): The participant will lie prone and the Placebo HILT will be administered is the same capacity as the treatment group however no Laser treatment will be administered. Upon conclusion of the placebo treatment, the skin with be evaluated for excessive redness or any other changes in skin appearance. Also, the participant will be asked about any discomfort.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: CureWave High Intensity Laser — * The participant will lie prone and the HILT will be administered in 9 symmetrical positions which cover the lumbosacral region. Dose will be 1minute per position. The dose will include:
    * Power (44 Watts)
    * Mode (continues wave)
    * Time on (60000 ms)
    * Time off (1 ms)
    * Repeats (9)
  * Distance of electrode from skin will begin 10" from skin surface. The participant may or may not feel mild warmth. Should the subject report excessive warmth or discomfort the probe distance will be increased in 2" intervals until it is comfortable. The entire process will take approximately 10 minutes.
  * The participant will lie prone and the Placebo treatment will consist of positioning the HILT probe over the 9 symmetrical positions for 1 minutes each however the no laser will be admitted.
  Arms: CureWave High Intensity Laser
Other: Placebo — The participant will lie prone and the NON ACTIVE HILT will be administered in 9 symmetrical positions which cover the lumbosacral region. Dose will be 1minute per position. THE LASER WILL NOT BE ACTIVE.
  o Distance of electrode from skin will begin 10" from skin surface. The entire process will take approximately 10 minutes.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effects of CureWave laser on paraspinal muscle oxygenation, pressure pain thresholds, muscle edema, and quality, and perceived outcomes in patients with chronic low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) contributes to disability and has a significant economic impact. High intensity laser devices are class 4 producing > 40 W of power at longer wavelengths, thereby allowing deeper tissue penetration. Currently, there is little evidence to demonstrate the effectiveness of high intensity laser treatment in those with chronic LBP. Optimal dosing strategies are still unknown as well as patient response based on chronicity of symptoms. Therefore, our study seeks to evaluate the effectives of high intensity laser therapy using CureWave in those with LBP of a duration longer than 3 months and with a dosing strategy of two times/week for three weeks.

Hypothesis

1. CureWave laser therapy will increase total oxygenated hemoglobin and muscle blood flow in patients with chronic LBP.
2. CureWave laser therapy will reduce inflammation as assessed by muscle edema in patients with chronic LBP.
3. CureWave laser therapy will improve paraspinal echogenicity (muscle quality) following treatment in patients with chronic LBP.
4. CureWave laser therapy will decrease muscle sensitivity in patients with chronic LBP
5. CureWave laser therapy will demonstrate improve patient reported outcomes, including decreased pain, reduced disability and improved function in patients with chronic LBP.
6. CureWave laser therapy will increase muscle activation during maximal strength testing.
7. CureWave laser therapy will decrease performance fatigability as assessed by maximal muscle activation and force production.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Self-reported history of low back pain (5 episodes in lifetime or 3 in last three years which altered activities of daily living)13

Exclusion Criteria:

* Self-reported pregnancy
* Inability to complete all required meeting sessions
* Known cardiovascular, pulmonary, metabolic, muscular, and/or coronary heart disease
* Regularly uses prescription medication
* Seeking medical care for the current episode of low back pain
* Report average symptoms greater than 8/10
* Inability to perceive light touch.
* Verbal reports of known cardiovascular, pulmonary, metabolic, muscular, and/or coronary heart disease
* Verbal reports of known skin sensitivity to gels or adhesives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
CHANGE in EMG activity of the lumbar paraspinal muscles | Baseline; 24-48 hours after baseline; 4 weeks after baseline
  EMG will be recorded during all submaximal and maximal strength testing. EMG will be assessed using wireless Bluetooth electrodes that will be attached using double-sided adhesive stickers. All submaximal and maximal strength testing will be performed using a hand-held dynamometer (Microfet 2 Manual Muscle Tester). Subjects will be stabilized using a nylon strap, the same material and mechanism as a seat belt, when necessary to eliminate accessory or compensatory motion during strength testing. This will be placed on their anterior and/or medial thigh with padding to eliminate any discomfort where the strap contacts the skin.
CHANGE in total hemoglobin | Baseline; 24-48 hours after baseline; 4 weeks after baseline
  Change in total hemoglobin will be used as an index of change in regional blood volume.will be assessed using near-infrared spectroscopy (NIRS) (Portamon, Artinis Medical Systems, Arnhem, The Netherlands).
CHANGE in Muscle Edema | Baseline; 24-48 hours after baseline; 4 weeks after baseline
  Muscle edema will be assessed via ultrasound using the echo intensity function. Ultrasound images will be obtained using a portable brightness mode (B-mode) ultrasound-imaging device (GE Logiqe, USA) and a multi-frequency linear-array probe (12L-Rs; 5-13MHz; 38.4 mm field-of-view). Ultrasound images will be analyzed using ImageJ software (Version 1.47v., National Institutes of Health, Bethesda, MD, USA). Echo intensity, as assessed by gray-scale analysis (0 arbitrary units [AU], corresponds to black image, 255 AU corresponds to white image) will be performed using the histogram function and will be determined from the same region of interest as muscle thickness.
CHANGE in Muscle sensitivity | Baseline; 24-48 hours after baseline; 4 weeks after baseline
  Muscle sensitivity will be measured with a handheld digital algometer (Wagner FDX-25 pressure algometer- Wagner Instruments, Greenwich, CT) and be applied at a right angle to the skin surface with the subject lying in prone position at 3 locations on the Paravertebral muscles, Quadratus lumborum, and Piriformis. Pressure will be applied at a rate of 30 kPa/s, which corresponds to 3 N/s.
CHANGE in Numeric Pain Rating Scale | Baseline; 24-48 hours after baseline; 4 weeks after baseline
  Quantity of perceived Pain will be evaluated via a likert scale between 0 (no pain) to 10 (the worst imaginable pain)
CHANGE in Muscle Oxygenation | Baseline; 24-48 hours after baseline; 4 weeks after baseline
  Muscle oxygenation will be assessed using near-infrared spectroscopy (NIRS) (Portamon, Artinis Medical Systems, Arnhem, The Netherlands). Changes in muscle tissue oxygenation and deoxyhemoglobin will be examined across time using the optical densities from two continuous wavelengths (760 and 850 nm)

SECONDARY OUTCOMES:
CHANGE in Oswestry Disability Index | Baseline; 24-48 hours after baseline; 4 weeks after baseline
  Measure self reported perceived disability via a standardized survey form that can report a raw score between 0 and 50 points.
CHANGE in Patients Specific Functional Scale | Baseline; 24-48 hours after baseline; 4 weeks after baseline
  Measure self reported functional abilities based on a survey form which identifies 5 individual functional tasks that the participant struggles with. These are rated 0 (no difficulty) to 10 (unable to perform task).
CHANGE in Global Rating of Change | Baseline; 24-48 hours after baseline; 4 weeks after baseline
  Measure overall change in condition via a survey questionnaire which rates change in symptoms between -7 (quite a bit worse) to 0 (no change) to +7 (quite a bit better).
CHANGE in Sleep disturbance (short form 8a) | Baseline; 24-48 hours after baseline; 4 weeks after baseline
  Measure self reported measures of sleep quality via a survey questionnaire that evaluates quality and quantity of sleep.
CHANGE in International Physical Activity Questionnaire (IPAQ) | Baseline; 24-48 hours after baseline; 4 weeks after baseline
  Measure of self reported physical activity via a survey questionnaire that reports level of physical activity.
CHANGE in McGill Pain Questionnaire | Baseline; 24-48 hours after baseline; 4 weeks after baseline
  Measure of pain quality via a survey questionnaire the measures qualitative aspects of perceived pain.

CONTACTS AND LOCATIONS:
Overall Officials: William J Hanney, PhD, Principal Investigator — University of Central Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Santamato A, Solfrizzi V, Panza F, Tondi G, Frisardi V, Leggin BG, Ranieri M, Fiore P. Short-term effects of high-intensity laser therapy versus ultrasound therapy in the treatment of people with subacromial impingement syndrome: a randomized clinical trial. Phys Ther. 2009 Jul;89(7):643-52. doi: 10.2522/ptj.20080139. Epub 2009 May 29. PMID 19482902
- [Background] Nakamura T, Ebihara S, Ohkuni I, Izukura H, Harada T, Ushigome N, Ohshiro T, Musha Y, Takahashi H, Tsuchiya K, Kubota A. Low Level Laser Therapy for chronic knee joint pain patients. Laser Ther. 2014 Dec 27;23(4):273-7. doi: 10.5978/islsm.14-OR-21. PMID 25705083
- [Background] Alghadir A, Omar MT, Al-Askar AB, Al-Muteri NK. Effect of low-level laser therapy in patients with chronic knee osteoarthritis: a single-blinded randomized clinical study. Lasers Med Sci. 2014 Mar;29(2):749-55. doi: 10.1007/s10103-013-1393-3. Epub 2013 Aug 3. PMID 23912778
- [Background] Fukuda VO, Fukuda TY, Guimaraes M, Shiwa S, de Lima Bdel C, Martins RA, Casarotto RA, Alfredo PP, Bjordal JM, Fucs PM. SHORT-TERM EFFICACY OF LOW-LEVEL LASER THERAPY IN PATIENTS WITH KNEE OSTEOARTHRITIS: A RANDOMIZED PLACEBO-CONTROLLED, DOUBLE-BLIND CLINICAL TRIAL. Rev Bras Ortop. 2015 Dec 6;46(5):526-33. doi: 10.1016/S2255-4971(15)30407-9. eCollection 2011 Sep-Oct. PMID 27027049
- [Background] Alayat MS, Elsodany AM, El Fiky AA. Efficacy of high and low level laser therapy in the treatment of Bell's palsy: a randomized double blind placebo-controlled trial. Lasers Med Sci. 2014 Jan;29(1):335-42. doi: 10.1007/s10103-013-1352-z. Epub 2013 May 26. PMID 23709010
- [Background] Kim SH, Kim YH, Lee HR, Choi YE. Short-term effects of high-intensity laser therapy on frozen shoulder: A prospective randomized control study. Man Ther. 2015 Dec;20(6):751-7. doi: 10.1016/j.math.2015.02.009. Epub 2015 Mar 2. PMID 25770420
- [Background] de Freitas LF, Hamblin MR. Proposed Mechanisms of Photobiomodulation or Low-Level Light Therapy. IEEE J Sel Top Quantum Electron. 2016 May-Jun;22(3):7000417. doi: 10.1109/JSTQE.2016.2561201. PMID 28070154
- [Background] Karlekar A, Bharati S, Saxena R, Mehta K. Assessment of feasibility and efficacy of Class IV laser therapy for postoperative pain relief in off-pump coronary artery bypass surgery patients: A pilot study. Ann Card Anaesth. 2015 Jul-Sep;18(3):317-22. doi: 10.4103/0971-9784.159800. PMID 26139735
- [Background] Chow R, Armati P, Laakso EL, Bjordal JM, Baxter GD. Inhibitory effects of laser irradiation on peripheral mammalian nerves and relevance to analgesic effects: a systematic review. Photomed Laser Surg. 2011 Jun;29(6):365-81. doi: 10.1089/pho.2010.2928. Epub 2011 Apr 1. PMID 21456946
- [Background] Basford JR, Sheffield CG, Harmsen WS. Laser therapy: a randomized, controlled trial of the effects of low-intensity Nd:YAG laser irradiation on musculoskeletal back pain. Arch Phys Med Rehabil. 1999 Jun;80(6):647-52. doi: 10.1016/s0003-9993(99)90167-3. PMID 10378490
- [Background] Ay S, Dogan SK, Evcik D. Is low-level laser therapy effective in acute or chronic low back pain? Clin Rheumatol. 2010 Aug;29(8):905-10. doi: 10.1007/s10067-010-1460-0. Epub 2010 Apr 23. PMID 20414695
- [Background] Fiore P, Panza F, Cassatella G, Russo A, Frisardi V, Solfrizzi V, Ranieri M, Di Teo L, Santamato A. Short-term effects of high-intensity laser therapy versus ultrasound therapy in the treatment of low back pain: a randomized controlled trial. Eur J Phys Rehabil Med. 2011 Sep;47(3):367-73. Epub 2011 Jun 8. PMID 21654616
- [Background] Hart JM, Fritz JM, Kerrigan DC, Saliba EN, Gansneder BM, Ingersoll CD. Quadriceps inhibition after repetitive lumbar extension exercise in persons with a history of low back pain. J Athl Train. 2006 Jul-Sep;41(3):264-9. PMID 17043693
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343

DOCUMENTS (1):
  • Informed Consent Form (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT04808492/ICF_000.pdf